CLINICAL TRIAL: NCT00677040
Title: Normal Tissue Oxygenation Following Radiotherapy
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Principal Investigator, Ken Dornfeld, Radiation Oncologist, Essentia Health
Other Study IDs: 030804
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-05

CONDITIONS: Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study involves women who have had a diagnosis of breast cancer, and have had a lumpectomy with radiation treatments completed in the past year.

The study will determine the level of oxygen in the skin of the breast that has been radiated, compared with the normal skin of the opposite breast.

The purpose of this study is to determine if there is a decrease in oxygen levels in the skin which has been radiated, hopefully to find a treatment to limit skin damage caused by radiation treatments, for women with breast cancer in the future.

DETAILED DESCRIPTION:
Successful completion of this study will provide data on changes in oxygenation in irradiated tissues. If changes are documented, this study would provide evidence supporting current models of tissue injury following radiotherapy. In addition, these data may provide a mechanistic rationale for clinical approaches to ameliorate the toxicities of radiotherapy. Finally, if a correlation exists between tissue oxygenation and toxicity, the rapid and simple tissue oxygenation test may provide a quantitative measure of toxicity and allow earlier and more precise assessment of both toxicity and efficacy of ameliorative therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast malignancy
2. Completion of breast irradiation one year (+/- 8 weeks) prior.
3. Surgical treatment with lumpectomy

Exclusion Criteria:

1. Inability to tolerate the 20 minute transcutaneous oxygenation measurements
2. Allergy to adhesives
3. Bilateral disease or absence of control breast or previous radiotherapy to "control" breast
4. More than one course of radiotherapy to the breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone breast conserving therapy consisting of lumpectomy and pPatients with breast cancer who received postoperative radiotherapy for breast conservation will be identified from tumor registry data and recruited into the study if they have completed radiotherapy less than one year ostoperative radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Dornfeld, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Background] Denham JW, Hauer-Jensen M. The radiotherapeutic injury--a complex 'wound'. Radiother Oncol. 2002 May;63(2):129-45. doi: 10.1016/s0167-8140(02)00060-9. PMID 12063002
- [Background] Archambeau JO, Pezner R, Wasserman T. Pathophysiology of irradiated skin and breast. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1171-85. doi: 10.1016/0360-3016(94)00423-I. PMID 7713781
- [Background] Brush J, Lipnick SL, Phillips T, Sitko J, McDonald JT, McBride WH. Molecular mechanisms of late normal tissue injury. Semin Radiat Oncol. 2007 Apr;17(2):121-30. doi: 10.1016/j.semradonc.2006.11.008. PMID 17395042
- [Background] Westbury CB, Pearson A, Nerurkar A, Reis-Filho JS, Steele D, Peckitt C, Sharp G, Yarnold JR. Hypoxia can be detected in irradiated normal human tissue: a study using the hypoxic marker pimonidazole hydrochloride. Br J Radiol. 2007 Nov;80(959):934-8. doi: 10.1259/bjr/25046649. Epub 2007 Oct 1. PMID 17908818
- [Background] Brizel DM, Wasserman TH, Henke M, Strnad V, Rudat V, Monnier A, Eschwege F, Zhang J, Russell L, Oster W, Sauer R. Phase III randomized trial of amifostine as a radioprotector in head and neck cancer. J Clin Oncol. 2000 Oct 1;18(19):3339-45. doi: 10.1200/JCO.2000.18.19.3339. PMID 11013273
- [Background] Delanian S, Depondt J, Lefaix JL. Major healing of refractory mandible osteoradionecrosis after treatment combining pentoxifylline and tocopherol: a phase II trial. Head Neck. 2005 Feb;27(2):114-23. doi: 10.1002/hed.20121. PMID 15641107
- [Background] Delanian S, Porcher R, Rudant J, Lefaix JL. Kinetics of response to long-term treatment combining pentoxifylline and tocopherol in patients with superficial radiation-induced fibrosis. J Clin Oncol. 2005 Dec 1;23(34):8570-9. doi: 10.1200/JCO.2005.02.4729. Epub 2005 Oct 31. PMID 16260695
- [Background] Bui QC, Lieber M, Withers HR, Corson K, van Rijnsoever M, Elsaleh H. The efficacy of hyperbaric oxygen therapy in the treatment of radiation-induced late side effects. Int J Radiat Oncol Biol Phys. 2004 Nov 1;60(3):871-8. doi: 10.1016/j.ijrobp.2004.04.019. PMID 15465205
- [Background] Marx RE, Johnson RP, Kline SN. Prevention of osteoradionecrosis: a randomized prospective clinical trial of hyperbaric oxygen versus penicillin. J Am Dent Assoc. 1985 Jul;111(1):49-54. doi: 10.14219/jada.archive.1985.0074. PMID 3897335
- [Background] Rudolph R, Tripuraneni P, Koziol JA, McKean-Matthews M, Frutos A. Normal transcutaneous oxygen pressure in skin after radiation therapy for cancer. Cancer. 1994 Dec 1;74(11):3063-70. doi: 10.1002/1097-0142(19941201)74:113.0.co;2-c. PMID 7880243
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Hauser CJ, Shoemaker WC. Use of a transcutaneous PO2 regional perfusion index to quantify tissue perfusion in peripheral vascular disease. Ann Surg. 1983 Mar;197(3):337-43. doi: 10.1097/00000658-198303000-00014. PMID 6830339
- [Background] Moore DS and McCabe GP. Introduction to the practice of statistics. New York: W.H. Freeman and Co., 2006.

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects: patients were invited to participate one year after completing radiotherapy as part of their treatment for breast preservation cancer treatment
Period: Overall Study
Arm/Group | Subjects
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 63 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants] — 20 female breast cancer patients were invited to participate one year after receiving radiation for part of their breast cancer treatment. Transcutaneous oxygen levels were measured for both breasts. Oxygen levels in the treated and non-treated breast were compared. The non treated breast levels serve as baseline levels.
  Participants
    Female | 20
    Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
tissue oxygenation of nontreated breast [Mean (Standard Deviation); unit: mmHg] — oxygenation was not measured prior to radiothearpy
  mmHg | 66.3 (22.8)

OUTCOME MEASURES:

1. Primary Outcome: Tissue Oxygenation
Description: Transcutaneous oxygen detector is used to measure the partial pressure of oxygen. The unit detects electrolytes ionized by oxygen. The measuring electrode also heats the skin being measured to facilitate maximal bloodflow to the area.
Time Frame: One visit for 20 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects
Number analyzed (Participants) | 20
mmHg | 62.5 (18.4)
Statistical Analysis 1: Comparison: Subjects; Test type: Equivalence — t-test to determine if tissue oxygen measurements are equivalent between treated and nontreated breast; p = 0.5, t-test, 2 sided; t-test = 0.35
Statistical Analysis 2: Comparison: Subjects; Test type: Other; p = .5, t-test, 2 sided; t-test = .35

2. Secondary Outcome: Skin and Soft Tissue Toxicity Will be Assessed Using the RTOG/EORTC Late Radiation Morbidity Scoring Schema When Oxygenation is Measured.
Time Frame: One visit
Measure: Count of Participants; unit: Participants
Groups:
- Subjects: patients were invited to participate one year after completing radiotherapy as part of their treatment for breast preservation cancer treatment. No adverse events were detected.
Arm/Group | Subjects
Number analyzed (Participants) | 20
Participants
  late subcutaneous toxicitiy score 1 | 19
  late subcutaneous toxcity score 2 | 1
  late skin toxicity score 1 | 19
  late skin toxicity score 2 | 1

ADVERSE EVENTS:
Description: no adverse events were found following the brief, 20 minute transcutaneous oxygen measurements
Arm/Group | Subjects
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes